CLINICAL TRIAL: NCT02683369
Title: Effects of a Commercially-available, Low-dose Iron Supplement (BloodBuilder®/Iron Response®) on Markers of Iron Status Among Premenopausal and Non-anemic, Iron-deficient Women
Brief Title: Low-dose Iron Supplementation and Markers of Iron Status Among Non-anemic, Iron-deficient Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Chris D'Adamo, Director of Research Center for Integrative Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 017-FS; HP-00067251
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Non-anemic Iron Deficiency
Keywords: Non-anemic Iron Deficiency, Iron Supplementation
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Iron Supplement (Experimental): Participants will consume one tablet of Blood Builder®/Iron Response®, once per day, every day, for 8 weeks.
  Interventions: Dietary Supplement: Blood Builder®/Iron Response®

INTERVENTIONS:
Dietary Supplement: Blood Builder®/Iron Response® — The low-dose iron dietary supplement is a tablet that contains vitamins and minerals selected to help maintain healthy red blood cells and iron levels in the blood. The supplement ingredients aim to generate a supplement by taking a food which contains the naturally occurring, complex matrix of proteins, lipids, carbohydrates and all other elements associated with the vitamin or mineral of interest. These natural food sources are used to generate tablets that maintain the vitamin and mineral potency found in the original food source as well as the associated elements that naturally accompany it.
  One tablet will be taken once a day offering a total daily serving of:
  * 15 mg of Vitamin C
  * 400 mcg of Folate
  * 30 mcg Vitamin of B-12
  * 26 mg of Iron
  * 125 mg of Beet Root
  Other Names: Low-dose iron dietary supplement

SUMMARY:
Healthy premenopausal women that are iron-deficient without anemia will receive a low-dose iron dietary supplement. The investigators seek to determine if the low-dose iron dietary supplement will restore iron levels to normal range with fewer side effects than typically experienced at higher doses of iron supplementation.

DETAILED DESCRIPTION:
The primary purpose of this clinical trial is to evaluate the impact of a low-dose iron dietary supplement on markers of iron status among a sample of premenopausal women that are iron-deficient without anemia. This study will also assess the incidence of mild adverse events (constipation, nausea, etc.) that are relatively common with other over the counter iron dietary supplements and that the investigators hypothesize will be reduced with this lower-dose formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal
2. Iron deficient without anemia (serum ferritin concentration < 20 ug/L and a hemoglobin concentration > 120 g/L)
3. Agree to continue with current diet and any dietary supplements
4. Able to understand and write English
5. Voluntarily consent to the study and understand its nature and purpose including potential risks and side effects

Exclusion Criteria:

1. Daily supplementation of another iron supplement (other than multivitamin) currently or within past 2 weeks
2. Pregnant or breastfeeding females
3. History of alcohol, drug, or medication abuse
4. Known allergies to any substance in the study product
5. Donated blood in the past month or plan to do so at any time during the 8-week trial
6. Current diagnosis of inflammatory bowel disease (Crohn's or Ulcerative Colitis)
7. Taking medication that my interfere with the absorption of iron
8. Current tobacco smoker

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-02; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Changes in Hemoglobin (Hgb) Level | Baseline and study end (8 weeks from baseline)
  Marker of iron status
Changes in Serum Ferritin (SF) Level | Baseline and study end (8 weeks from baseline)
  Marker of iron status
Changes in Soluble Transferrin Receptor (sTfR) Level | Baseline and study end (8 weeks from baseline)
  Marker of iron status
Changes in Total Body Iron Stores | Baseline and study end (8 weeks from baseline)
  Marker of iron status

SECONDARY OUTCOMES:
Frequency and severity of self-reported constipation | Study end (8 weeks from baseline)
Frequency and severity of self-reported diarrhea | Study end (8 weeks from baseline)
Frequency and severity of self-reported nausea | Study end (8 weeks from baseline)
Frequency and severity of self-reported vomiting | Study end (8 weeks from baseline)
Frequency and severity of self-reported fatigue | Baseline and study end (8 weeks from baseline)
Self-reported energy level | Baseline and study end (8 weeks from baseline)
Supplement compliance assessed using participant daily diary | Study end (8 weeks from baseline)
Adverse events | Study end (8 weeks from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Chris D'Adamo, PhD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Center for Integrative Medicine University of Maryland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Adamo CR, Novick JS, Feinberg TM, Dawson VJ, Miller LE. A Food-Derived Dietary Supplement Containing a Low Dose of Iron Improved Markers of Iron Status Among Nonanemic Iron-Deficient Women. J Am Coll Nutr. 2018 May-Jun;37(4):342-349. doi: 10.1080/07315724.2018.1427158. Epub 2018 Mar 13. PMID 29533710